CLINICAL TRIAL: NCT06373159
Title: A Study for the Disseminated Intravascular Coagulation Among Patients With Sepsis in Japan: A Hospital-based Cohort Study
Brief Title: An Observational Study to Learn About the Occurrence of Disseminated Intravascular Coagulation Among Adults With Sepsis in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22643
Record Dates: First submitted 2024-03-25; First posted 2024-04-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Disseminated Intravascular Coagulation
Keywords: Thrombocytopenic sepsis; Septic shock
MeSH Terms: conditions — Sepsis; Disseminated Intravascular Coagulation; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sepsis patient cohort: Patients diagnosed with sepsis in patient inclusion period, regardless of etiology, including subgroups: sepsis with thrombocytopenia patient cohort and septic shock patient cohort
  Interventions: Other: No study intervention
- Sepsis-associated DIC patient cohort: Sepsis patients with onset of DIC in the patient record in patient inclusion period
  Interventions: Other: No study intervention
- Non-sepsis-associated DIC patient cohort: DIC patients without sepsis in patient inclusion period
  Interventions: Other: No study intervention

INTERVENTIONS:
Other: No study intervention — Retrospective observational study using Real World Data (RWD) in Japan without study intervention

SUMMARY:
This is an observational study in which data already collected from people with sepsis (blood poisoning) and/or disseminated intravascular coagulation (DIC) are studied.

In observational studies, only observations are made without participants receiving any advice or changes to their healthcare.

DIC is a serious blood disorder that can cause clots throughout the body, blocking blood vessels. People who have sepsis or cancer are at a higher risk of developing DIC.

To find a treatment that works well for people with DIC associated with sepsis, it is important to know about its occurrence, treatments people receive, and their outcomes. Japan is the only country that has officially approved medicines for DIC including a few newer medicines that prevent extensive blood clotting.

In this study, researchers will assess patient data from a hospital database in Japan.

The main purpose of this study is to learn more about how many adults develop DIC related to sepsis, thrombocytopenic sepsis (sudden decrease in the number of platelets in the blood), or septic shock (dangerously low blood pressure) in Japan every year.

To learn about this, researchers will collect the following information:

* The number of participants who developed DIC 14 days, 21 days and 28 days after their sepsis diagnosis
* The grading scores given to the participants which are used to assess the likelihood, cause, severity, treatment plan, and outcome of DIC (including scores called JAAM, ISTH, MHLW, and/or SOFA scores)
* The number of days between diagnosis of sepsis and the beginning of DIC

Researchers will study the data collected between June 2018 and June 2023. The data will come from TXP Medical, which collects data through the hospital health information system of 7 selected hospitals for this study across Japan.

In this study, only available data from routine care are collected.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis patient cohort

  * Sepsis patients
  * Age ≥18 years
  * Subgroups:

    * Sepsis with thrombocytopenia patient cohort
    * Septic shock patient cohort
* Sepsis-associated DIC patient cohort

  * DIC patients in sepsis patient cohort
  * Subgroups:

    * Organ failure: kidney (Serum creatinine (SCr) < 1.2 mg/dl and ≥ 1.2 mg/dl)
    * Organ failure: liver (bilirubin < 1.2 mg/dl and ≥ 1.2 mg/dl)
    * Organ failure: cardiovascular (with and without catecholamine or vasopressin)
    * With low molecular weight (LMW) heparins, unfractionated heparins, and both
    * With and without DIC treatment

      * Priority 1_Anticoagulants specifically used in Japan (recombinant antithrombin, recombinant thrombomodulin, human anti-thrombin III)
      * Priority 1 + Priority 2_Drugs for sepsis-associated DIC (LMW heparins, unfractionated heparins, protease inhibitors)
      * Priority 1 + Priority 2 + Priority 3_antibiotics (antifungals), and/or steroids
* Non-sepsis-associated DIC patient cohort

  * Hematopoietic malignant tumor patients
  * DIC patients
  * Age ≥18 years

Exclusion Criteria:

* Sepsis patient cohort: None
* Sepsis-associated DIC patient cohort: None
* Non-sepsis-associated DIC patient cohort: Sepsis patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Source population are patients in hospitals providing electronic medical record (EMR) and diagnosis procedure combination (DPC) data to TXP Medical in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 5740 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Incidence of DIC assessed at 14 days, 21 days and 28 days of the patient follow up | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  DIC: disseminated intravascular coagulation
Distribution of JAAM DIC score | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  The Japanese Association for Acute Medicine (JAAM) DIC scoring algorithm includes a number of variables but in addition specific criteria for evidence of a Systemic Inflammatory Response Syndrome (SIRS). JAAM DIC score >= 4 supports a diagnosis of DIC. DIC: disseminated intravascular coagulation
Distribution of ISTH DIC score | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  The International Society on Thrombosis Haemostasis (ISTH) DIC score is a simple scoring system produced by the ISTH group for the diagnosis of DIC depending on the Platelet count, the PT, the fibrinogen level and critically the FDP/D-Dimer results. A total score of ≥5 = DIC as long as the score is associated with a clinical disorder known to cause DIC. DIC: disseminated intravascular coagulation
Distribution of MHLW DIC score | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  The Japanese Ministry of Health, Labor and Welfare (MHLW) DIC score is a scoring system for the diagnosis of overt DIC. MHLW DIC score ≥7 is defined as DIC. DIC: disseminated intravascular coagulation
Distribution of SOFA score | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  The Sequential Organ Failure Assessment (SOFA) score is a scoring system based on performance of respiratory, coagulation, liver, cardiovascular, central nervous system, and kidney. The higher the SOFA score, the higher the likely mortality. DIC: disseminated intravascular coagulation
Days from sepsis diagnosis to the onset of DIC | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  DIC: disseminated intravascular coagulation

SECONDARY OUTCOMES:
Number of participants per clinical characteristics | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  Clinical characteristics (e.g., demographics, comorbidities, medical history) in patients with sepsis, thrombocytopenic sepsis and septic shock, respectively; in patients with sepsis in different definitions (diagnosis codes, laboratory values, and procedure codes); at the onset of DIC in patients who developed sepsis-associated DIC. DIC: disseminated intravascular coagulation
Number of participants per DIC treatment patterns in patients with sepsis-associated DIC following the onset of DIC | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  DIC: disseminated intravascular coagulation
Incidence rates of clinical outcomes assessed in patients with sepsis-associated DIC | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  Clinical outcomes are assessed at 14 days, 28 days, 60 days, 183 days, 365 days (1 year) and 730 days (2 years) of follow up. Clinical outcomes include thrombosis, major bleeding, organ failures, death, ICUs admission during the index hospitalization, discharge during the index hospitalization, length of index hospitalization. DIC: disseminated intravascular coagulation
Cumulative incidences of clinical outcomes assessed in patients with sepsis-associated DIC | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  Clinical outcomes are assessed at 14 days, 28 days, 60 days, 183 days, 365 days (1 year) and 730 days (2 years) of follow up. Clinical outcomes include thrombosis, major bleeding, organ failures, death, ICUs admission during the index hospitalization, discharge during the index hospitalization, length of index hospitalization. DIC: disseminated intravascular coagulation
Number of participants per clinical characteristics in subgroup of patients who developed sepsis-associated DIC | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  DIC: disseminated intravascular coagulation
Number of participants per treatment patterns in subgroup of patients who developed sepsis-associated DIC | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  DIC: disseminated intravascular coagulation
Incidence rates of clinical outcomes in subgroup of patients who developed sepsis-associated DIC | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  Clinical outcomes include thrombosis, major bleeding, organ failures, death, ICUs admission during the index hospitalization, discharge during the index hospitalization, length of index hospitalization.
Number of participants per clinical characteristics after the onset of DIC in patients with non-sepsis-associated DIC | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  DIC: disseminated intravascular coagulation
Number of participants per treatment patterns after the onset of DIC in patients with non-sepsis-associated DIC | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  DIC: disseminated intravascular coagulation
Incidence rates of clinical outcomes after the onset of DIC in patients with non-sepsis-associated DIC | Retrospective analysis of real world data between 01 JUN 2018 and 01 JUN 2023
  Clinical outcomes include thrombosis, major bleeding, organ failures, death, ICUs admission during the index hospitalization, discharge during the index hospitalization, length of index hospitalization.

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.